CLINICAL TRIAL: NCT03727516
Title: Validation of the Cross-cultural Adapted Italian Version of the Oxford Elbow Score
Brief Title: Italian Version of the Oxford Elbow Score Score
Acronym: Italian-OES
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Sara Padovani, Medical Doctor, Principal Investigator, Orthopaedic Resident, Università degli Studi di Ferrara
Other Study IDs: 95/2018/Oss/AOUFe
Record Dates: First submitted 2018-10-22; First posted 2018-11-01 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Elbow Disease; Patients Reported Outcomes; Elbow Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergone elbow surgery: Patients undergone elbow surgery at routine follow up at 2 or 6 months

SUMMARY:
Validation of the cross-cultural adapted Italian version of the Oxford Elbow Score, in order to have an instrument able to detect the functional state reported by patients after elbow surgery.

DETAILED DESCRIPTION:
An Italian version of the Oxford Elbow Score has been created by an experts committee, according to the published guidelines for the cross-cultural adaptation of self-reported measures.

The new version of the questionnaire will be administered to a sample size of 120 patients, in addition to MEPS, Quick DASH and SF-36 questionnaires during the follow-up apointments at 2 and/or 6 months after elbow surgery in two Orthopaedic Clinic in North Italy.

Reliability, validity , reproducibility and responsiveness will be detected by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak and understand Italian,
* need for one-elbow surgical procedure any elbow disease.

Exclusion Criteria:

* Injury in more than one musculoskeletal district

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is required a sample of 120 consecutive patients interviewed at routine follow up visit at 2 and/or 6 month after elbow surgery.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
the Italian version of the Oxford Elbow Score (OES) | up to 1 month post-surgery
  The Oxford Elbow Score (OES) is a disease-specific questionnaire, completed by patients, which assesses: pain, function and psychological status related to the elbow joint. Each domain is transformed into a 100-point score, where the highest value indicates a better condition. The total score is the result of the average of the three domains.
The Mayo Elbow Performance Score (MEPS) | up to 1 month post-surgery
  This questionnaire evaluates pain, range of motion, joint stability and the ability to perform 5 movements, respectively.
  The function of the elbow is considered excellent (score ≥ 90), good (75-89), modest (60-74), and poor (<60).
Quick Disability of Arm Shoulder and Hand | up to 1 month post surgery
  The Quick DASH is scored in two components: the disability/symptom section (11 items, scored 1-5) and the optional high performance sport/music or work modules (4 items, scored 1-5).
The Short Form - 36 (SF-36) Questionnaire | up to 1 month post-surgery
  The Sort Form-36 is widely used questionnaire to survey health related quality of life. The questionnaire is a 36-items that measures eight domains of health reporting a score from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Minimal clinical change of the Italian version of the Oxford El bow Score | Att 1month and 3 month post-surgery
  A group of patients will be interviewed at two different times points interval

CONTACTS AND LOCATIONS:
Overall Officials: Sara Padovani, M.D., Principal Investigator — Università degli Studi di Ferrara; Leo Massari, Study Chair — Università degli Studi di Ferrara
Locations (2):
- Italy (2):
  - Ospedale Degli Infermi di Faenza, Faenza, Ravenna
  - Azienda Ospedaliero-Universitaria Sant'Anna Cona, Ferrara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roquelaure Y, Ha C, Leclerc A, Touranchet A, Sauteron M, Melchior M, Imbernon E, Goldberg M. Epidemiologic surveillance of upper-extremity musculoskeletal disorders in the working population. Arthritis Rheum. 2006 Oct 15;55(5):765-78. doi: 10.1002/art.22222. PMID 17013824
- [Result] Vincent JI, MacDermid JC, King GJ, Grewal R. Validity and sensitivity to change of patient-reported pain and disability measures for elbow pathologies. J Orthop Sports Phys Ther. 2013 Apr;43(4):263-74. doi: 10.2519/jospt.2013.4029. Epub 2013 Mar 13. PMID 23485685
- [Result] Longo UG, Franceschi F, Loppini M, Maffulli N, Denaro V. Rating systems for evaluation of the elbow. Br Med Bull. 2008;87:131-61. doi: 10.1093/bmb/ldn023. Epub 2008 Jun 6. PMID 18539627
- [Result] Gummesson C, Atroshi I, Ekdahl C. The disabilities of the arm, shoulder and hand (DASH) outcome questionnaire: longitudinal construct validity and measuring self-rated health change after surgery. BMC Musculoskelet Disord. 2003 Jun 16;4:11. doi: 10.1186/1471-2474-4-11. Epub 2003 Jun 16. PMID 12809562
- [Result] Dawson J, Doll H, Boller I, Fitzpatrick R, Little C, Rees J, Jenkinson C, Carr AJ. The development and validation of a patient-reported questionnaire to assess outcomes of elbow surgery. J Bone Joint Surg Br. 2008 Apr;90(4):466-73. doi: 10.1302/0301-620X.90B4.20290. PMID 18378921
- [Result] Iordens GIT, Den Hartog D, Tuinebreijer WE, Eygendaal D, Schep NWL, Verhofstad MHJ, Van Lieshout EMM; FuncSiE Trial Investigators. Minimal important change and other measurement properties of the Oxford Elbow Score and the Quick Disabilities of the Arm, Shoulder, and Hand in patients with a simple elbow dislocation; validation study alongside the multicenter FuncSiE trial. PLoS One. 2017 Sep 8;12(9):e0182557. doi: 10.1371/journal.pone.0182557. eCollection 2017. PMID 28886018